CLINICAL TRIAL: NCT02982304
Title: Multi-Target Pallidal and Thalamic Deep Brain Stimulation for Hemi-Dystonia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H14-03185
Record Dates: First submitted 2016-11-14; First posted 2016-12-05 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Dystonia; Dystonia, Secondary
MeSH Terms: conditions — Dystonia; Dystonic Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pallidal (GPi) Deep Brain Stimulation (Active Comparator): GPi is the standard target for treating most dystonia. This setting will be the active comparator
  Interventions: Device: Deep Brain Stimulation
- Thalamic (Vim) Deep Brain Stimulation (Experimental): Vim is the standard target to treat cerebellar dysfunction in movement disorders. It is not routinely used in secondary dystonia
  Interventions: Device: Deep Brain Stimulation
- GPi + Vim (Multi-Target) Deep Brain Stimulation (Experimental): Combined stimulation of GPi and Vim stimulation (both electrodes ON)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation Electrode

SUMMARY:
Dystonia is increasingly being considered as a multi-nodal network disorder involving both basal ganglia and cerebellar dysfunction. The aim of this study is to determine if "Multi-Target" Thalamic and Pallidal Deep Brain Stimulation improves hemi-dystonia patients who are receiving inadequate therapy from GPi DBS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hemi-dystonia secondary to stroke
2. Candidate for GPi DBS
3. Able to provide informed consent

Exclusion Criteria:

1. History of intracranial pathology (such as multiple sclerosis, tumors, or aneurysms) that may account for dystonia or essential tremor.
2. History or evidence of ongoing psychiatric or neurodegenerative disorders (such as Parkinson's disease, Alzheimer's disease).
3. Incompetent adults or those unable to communicate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Burke Fahn Marsden Disability Rating Scale (BFMDRS) | 3 months
SF-36 Quality of Life Scale | 3 months
Adverse effects of Vim or Vim + GPi Neuromodulation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Honey, MD,DPhil,FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Slotty PJ, Poologaindran A, Honey CR. A prospective, randomized, blinded assessment of multitarget thalamic and pallidal deep brain stimulation in a case of hemidystonia. Clin Neurol Neurosurg. 2015 Nov;138:16-9. doi: 10.1016/j.clineuro.2015.07.012. Epub 2015 Jul 29. PMID 26241157
- [Background] Prudente CN, Hess EJ, Jinnah HA. Dystonia as a network disorder: what is the role of the cerebellum? Neuroscience. 2014 Feb 28;260:23-35. doi: 10.1016/j.neuroscience.2013.11.062. Epub 2013 Dec 11. PMID 24333801